CLINICAL TRIAL: NCT00566969
Title: Cocaine Withdrawal and Pharmacotherapy Response
Acronym: Carvedilol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0704002562; R01DA014537 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Cocaine Dependence; Opiate Dependence
Keywords: cocaine, opiate, methadone, carvedilol
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Sugars; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar Pill (Placebo Comparator): To be compared to active drug
  Interventions: Drug: sugar pill
- Carvedilol 25 mg (Active Comparator): To be compared to placebo and Carvedilol 50 mg
  Interventions: Drug: Carvedilol 25 mg
- Carvedilol 50 mg (Active Comparator): To be compared to placebo and Carvedilol 25 mg
  Interventions: Drug: Carvedilol 50 mg

INTERVENTIONS:
Drug: sugar pill — Subjects randomized to placebo, carvedilol 25mg or 50mg
  Other Names: placebo
  Arms: Sugar Pill
Drug: Carvedilol 25 mg — subjects randomized to placebo, carvedilol 25mg or 50mg
  Other Names: Coreg
  Arms: Carvedilol 25 mg
Drug: Carvedilol 50 mg — subjects randomized to placebo, carvedilol 25mg or 50mg
  Other Names: Coreg
  Arms: Carvedilol 50 mg

SUMMARY:
A total of 120 male and female opioid dependent cocaine users will participate in this study. This study will be a 8-week double-blind, placebo controlled study examining the dose-dependent effects of carvedilol (up to 50 mg/day) in methadone stabilized patients. The design will have two phases: 1) a four-week "treatment " phase; and 2) a 4 week " taper and detoxification or transfer" phase. Subjects will be cocaine users who are on stable doses of methadone (60 to 140 mg/day). Carvedilol dose will be increased from 12.5mg/day to the target dose of either 25 or 50 mg/day as tolerated. At the end of the treatment-phase, subjects will undergo detoxification from methadone over a 2 to 4-week period based on an individual's needs, and they will concurrently be tapered off carvedilol.

DETAILED DESCRIPTION:
The adrenergic neurotransmission serves multiple functions including learning, emotional processing and stress response to psychological and physical challenges (Huether, 1996; Sved et al., 2001). Adrenergic transmission also mediates drug withdrawal states and stress-induced relapse to drug use (Aston-Jones et al., 2004; Stewart, 2000). Consistent with these preclinical findings, adrenergic blockers showed promise as a treatment of cocaine dependence (Kampman et al., 2001b; Kampman et al., 2006). These preliminary findings are significant because there are no proven pharmacotherapies for cocaine addiction although an estimated 2.3 million of Americans aged 12 or older are regular cocaine users (SAMHSA, 2004). The societal cost of cocaine addiction is estimated to be $45 billion in the US, suggesting that development of even modestly effective cocaine pharmacotherapies will have great economic benefits. For example, availability of a medication decreasing cocaine use by 10 percent is estimated to have $745 million economic benefit in the US alone (Cartwright, 2000). Thus, developing effective treatments for cocaine addiction is an essential goal with significant benefits both for the society and the individual.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence as evidenced by documented prior treatment for opioid dependence or signs of opiate withdrawals, self-reported history of opioid dependence for a consecutive 12 month period and a positive urine for opiates.
* Current cocaine use with self-reported use of cocaine > 1 time/week in at least on month preceding study entry, provision of a cocaine-positive urine and fulfilled DSM-IV criteria for cocaine dependence
* For women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests.

Exclusion Criteria:

* current diagnosis of other drug or alcohol dependence (other than opiates, cocaine or tobacco);
* serious medical illness including asthma, diabetes, bradycardia, or other arrhythmias and major cardiovascular, renal, endocrine, hepatic disorders;
* current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder or significant current suicidal or homicidal thoughts;
* screening liver function tests (AST or ALT) greater than 3 times normal;
* known allergy or intolerance for carvedilol or methadone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: To be compared to active drug
  sugar pill: randomly given 25mg or 50mg of a sugar pill or the active comparator
- Carvedilol 25 mg; Carvedilol 50 mg: To be compared to sugar pill
  carvedilol: randomly assigned to 25mg or 50mg of Carvedilol or sugar pill, dose determined by height and weight.
Period: Overall Study
Arm/Group | Sugar Pill | Carvedilol 25 mg | Carvedilol 50 mg
Started | 34 | 37 | 35
Completed | 19 | 28 | 23
Not Completed | 15 | 9 | 12

BASELINE CHARACTERISTICS:
Population: 106 subjects meeting inclusion criteria who were without exclusions and randomized to an intervention.
Groups:
- Carvedilol 25 mg: To be compared to placebo and Carvedilol 50 mg
  carvedilol: subjects randomized to placebo, carvedilol 25mg or 50mg
- Carvedilol 50 mg: To be compared to placebo and Carvedilol 25 mg
  Carvedilol: subjects randomized to placebo, carvedilol 25mg or 50mg
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Carvedilol 25 mg | Carvedilol 50 mg | Total
Number analyzed (Participants) | 34 | 37 | 35 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (9.1) | 37.7 (10.9) | 39.1 (10.9) | 38.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 11 | 40
  Male | 19 | 23 | 24 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 10 | 4 | 26
  White | 21 | 24 | 25 | 70
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Abstinent From Cocaine - Self Report
Description: Percent Self reported days of abstinence from any cocaine use during the 11 week trial.
Time Frame: 11 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Sugar Pill | Carvedilol 25 mg | Carvedilol 50 mg
Number analyzed (Participants) | 19 | 28 | 23
percentage of days | 72.9 (25.3) | 72.9 (29) | 59.3 (31.7)
Statistical Analysis 1: Comparison: Sugar Pill vs Carvedilol 25 mg vs Carvedilol 50 mg; Test type: Non-Inferiority or Equivalence — A hierarchical linear model was used to account for unequal variance and covariance structures across time; p = .10, ANOVA

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Sugar Pill | Carvedilol 25 mg | Carvedilol 50 mg
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 14/19 | 13/28 | 13/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=19) | Carvedilol 25 mg (N=28) | Carvedilol 50 mg (N=23)
Disturbed concentration (Psychiatric disorders) | 6 (6) | 5 (5) | 7 (7)
Agitation (Psychiatric disorders) | 11 (11) | 13 (13) | 7 (7)
Tiredness (Psychiatric disorders) | 13 (13) | 13 (13) | 11 (11)
Drowsiness (Psychiatric disorders) | 6 (6) | 10 (10) | 7 (7)
Insomnia (Psychiatric disorders) | 14 (14) | 13 (13) | 11 (11)
Nightmares (Psychiatric disorders) | 5 (5) | 5 (5) | 7 (7)
Depression (Psychiatric disorders) | 10 (10) | 11 (11) | 11 (11)
Anxiety (Psychiatric disorders) | 8 (8) | 10 (10) | 11 (11)
Numbness (Nervous system disorders) | 3 (3) | 7 (7) | 7 (7)
Cramps (Nervous system disorders) | 4 (4) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 7 (7) | 9 (9) | 8 (8)
Constipation (Gastrointestinal disorders) | 13 (13) | 11 (11) | 13 (13)
Decreased appetitie (Gastrointestinal disorders) | 6 (6) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No